CLINICAL TRIAL: NCT01835600
Title: Suspension of Mechanical Ventilation in Ureteroscopic Lithotripsy Under General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Yi Zhou, Department of Anesthesiology , Changhai Hospital Affiliated to Second Military Medical, Chinese Medical Association
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SMV-312
Record Dates: First submitted 2013-04-02; First posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Hypercapnia; Hypoxia
MeSH Terms: conditions — Hypercapnia; Hypoxia | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with PEEP (Active Comparator): 10 cmH2O PEEP added to the respiratory curcuit during suspension of mechanical ventilation
  Interventions: Other: PEEP
- without PEEP (Placebo Comparator): 0 cmH2O PEEP added to the respiratory curcuit during suspension of mechanical ventilation

INTERVENTIONS:
Other: PEEP — PEEP means that when mechanical ventilation is suspended, the value of expiratory valve in the anesthesia machine is set at 10 cmH2O with 1 L/min 100% oxygen.
  Other Names: positive end-expiratory pressure
  Arms: with PEEP

SUMMARY:
For some upper ureteral and renal stones,ureteroscopic lithotripsy needs to be performed under general anesthesia with interrupted suspension of mechanical ventilation, which could result in hypercapnia and hypoxia. In this study, the investigators hypothesize that 10 cmH2O PEEP added to the respiratory circuit with 1 L/min 100% oxygen might extend the time of ventilation suspension but have no effect on carbon dioxide retention in blood.

DETAILED DESCRIPTION:
For some upper ureteral and renal stones,ureteroscopic lithotripsy is often perdurbed by the patient's respiratory movement either under epidural anesthesia or general anesthesia with mechanical ventilation. So intermittent suspension of mechanical ventilation under general anesthesia can ensure the surgery to be performed continuously and successfully. But this could result in hypercapnia and hypoxia. So far, there have been few studies focused on the change of the internal environment in blood as result of suspending breath. In this study, the investigators hypothesize that 10 cmH2O PEEP added to the respiratory circuit with 1 L/min 100% oxygen might extend the time of ventilation suspension but have no effect on carbon dioxide retention in blood.

ELIGIBILITY:
Inclusion Criteria:

ASA I~III general anesthesia sign the informed consent

Exclusion Criteria:

ASA IV or V woman who is pregnant or plans to bear

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-09 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
change in blood gas | Baseline before suspension of ventilation, 5 min after suspension, 10 min after suspension, 15 min after suspension, 5 min after re-ventilaiton, 10 min after re-ventilation
  we chose different time points to mesure the changes in blood gas.

SECONDARY OUTCOMES:
Change in systolic blood pressure | Baseline before suspension of ventilation, 5 min after suspension, 10 min after suspension, 15 min after suspension, 5 min after re-ventilaiton, 10 min after re-ventilation
  we chose different time points to mesure the changes in systolic blood pressure

OTHER OUTCOMES:
duration of the operation | from the start of the surgery to the end of the surgery
  We record the duration of the operation
recovery time | from the end of anesthesia to return of consciousness
  We record how long it will take for the patients to act accoreding to our order after ceasing anesthesia.
intraoperative awareness | from the initiation of anesthesia to the end of the surgery
  We will record if patinets have any memory during the operative, namely intraoperatiove awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Yi Zhou, Shanghai, Shanghai Municipality, China